CLINICAL TRIAL: NCT06963502
Title: A Phase Ib Study Evaluating the Safety, Tolerability , Pharmacokinetics，Activity and Immunogenicity of HS-10370 in Addition to Other Anti-cancer Therapies in Patients With Advanced Solid Tumors
Brief Title: A Phase Ib Study of HS-10370 in Addition to Other Anti-cancer Therapies in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-10370-103
Record Dates: First submitted 2025-04-16; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumors; Colorectal Cancer; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Capecitabine; Oxaliplatin; Leucovorin; Fluorouracil; Irinotecan; Platinum; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Arm 1:HS-10370 dose 1+ HS-20117 dose 3 (Experimental)
  Interventions: Drug: HS-10370; Drug: HS-20117
- Arm 2: HS-10370 dose 2 +HS-20117 dose 4+ Adebrelimab (Experimental)
  Interventions: Drug: HS-10370; Drug: HS-20117; Drug: Adebrelimab
- Arm 3: HS-10370 dose 1 + HS-20117 dose4 + Chemotherapy (Experimental)
  Interventions: Drug: HS-10370; Drug: HS-20117; Drug: Capecitabine; Drug: Oxaliplatin
- Arm 4: HS-10370 dose 1 + HS-20117 dose3 + Chemotherapy (Experimental)
  Interventions: Drug: HS-10370; Drug: HS-20117; Drug: Folinic Acid, Fluorouracil and Oxaliplatin/Irinotecan
- Arm 5:HS-10370 dose1+ HS-20117 dose 4+HS-20093 dose 5 (Experimental)
  Interventions: Drug: HS-10370; Drug: HS-20117; Drug: HS-20093
- Arm 6:HS-10370 dose 2 +HS-20093 dose 5+ Adebrelimab (Experimental)
  Interventions: Drug: HS-10370; Drug: Adebrelimab; Drug: HS-20093
- Arm 7:HS-10370 dose 2 +HS-20093 dose 6+ Adebrelimab+ Chemotherapy (Experimental)
  Interventions: Drug: HS-10370; Drug: Adebrelimab; Drug: HS-20093; Drug: platinum (cisplatin or carboplatin)

INTERVENTIONS:
Drug: HS-10370 — Participants will receive HS-10370 dose 1 administered orally
Drug: HS-20117 — Participants will receive HS-20117 given as dose 3 intravenous infusion(IV) once every 14-day cycle.
  Arms: Arm 1:HS-10370 dose 1+ HS-20117 dose 3; Arm 2: HS-10370 dose 2 +HS-20117 dose 4+ Adebrelimab; Arm 3: HS-10370 dose 1 + HS-20117 dose4 + Chemotherapy; Arm 4: HS-10370 dose 1 + HS-20117 dose3 + Chemotherapy; Arm 5:HS-10370 dose1+ HS-20117 dose 4+HS-20093 dose 5
Drug: Adebrelimab — Participants will receive Adebrelimab intravenous infusion(IV) once every 21-day cycle
  Arms: Arm 2: HS-10370 dose 2 +HS-20117 dose 4+ Adebrelimab; Arm 6:HS-10370 dose 2 +HS-20093 dose 5+ Adebrelimab; Arm 7:HS-10370 dose 2 +HS-20093 dose 6+ Adebrelimab+ Chemotherapy
Drug: Capecitabine — Participants will receive Capecitabine administered orally
  Arms: Arm 3: HS-10370 dose 1 + HS-20117 dose4 + Chemotherapy
Drug: Oxaliplatin — Participants will receive Oxaliplatin intravenous infusion(IV) once every 21-day cycle.
  Arms: Arm 3: HS-10370 dose 1 + HS-20117 dose4 + Chemotherapy
Drug: Folinic Acid, Fluorouracil and Oxaliplatin/Irinotecan — Participants will receive Folinic Acid, Fluorouracil and Oxaliplatin/Irinotecan intravenous infusion(IV) once every 14-day cycle.
  Arms: Arm 4: HS-10370 dose 1 + HS-20117 dose3 + Chemotherapy
Drug: HS-20093 — Participants will receive HS-20093 intravenous infusion(IV) once every 21-day cycle
  Arms: Arm 5:HS-10370 dose1+ HS-20117 dose 4+HS-20093 dose 5; Arm 6:HS-10370 dose 2 +HS-20093 dose 5+ Adebrelimab; Arm 7:HS-10370 dose 2 +HS-20093 dose 6+ Adebrelimab+ Chemotherapy
Drug: platinum (cisplatin or carboplatin) — Participants will receive platinum (cisplatin or carboplatin) administered IV in 21-day cycles.
  Arms: Arm 7:HS-10370 dose 2 +HS-20093 dose 6+ Adebrelimab+ Chemotherapy

SUMMARY:
This is a Phase Ib study that will evaluate the Safety, Tolerability , Pharmacokinetics, Activity and Immunogenicity of HS-10370 in Combination With Other Anti-cancer Therapies in Chinese patients with KRAS G12C mutation advanced or metastatic solid tumors, especially in and Colorectal cancer(CRC) and non-Small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Men or women greater than or equal to 18 years
* At least one measurable lesion in accordance with RECIST 1.1
* Must have an ECOG performance status of 0 or 1.
* Patients with advanced solid tumors who have failed after adequate standard treatment, are intolerant to standard treatment, or have no standard treatment available.
* Documentation of the presence of a KRAS G12C mutation
* Estimated life expectancy ≥12 weeks.
* Reproductive-age women agree to use adequate contraception and cannot breastfeed while participating in this study and for a period of 6 months after the last dose.Men also consent to use adequate contraceptive method within the same time limit.
* The subjects are able to comply with the process of the protocol.

Exclusion Criteria:

* Treatment with any of the following: Previous or current treatment with other KRAS G12C inhibitors.
* Active brain metastases.
* Patients with uncontrolled pleural, ascites or pericardial effusion
* Spinal cord compression
* Presence of Grade ≥ 2 toxicities due to prior anti-tumor therapy.
* Subjects with tumors known to harbor molecular alterations for which targeted therapy is locally approved, except for KRAS G12C.
* History of other primary malignancies.
* Inadequate bone marrow reserve or organ functions.
* Abnormal cardiac examination results.
* Severe, uncontrolled or active cardiovascular disorders.
* Diabetes ketoacidosis or hyperglycemia hyperosmolality
* Uncontrolled hypertension.
* Severe bleeding symptoms or bleeding tendencies.
* Severe arteriovenous thrombosis occurred
* Serious infection.
* Continuous use of glucocorticoids
* Active infectious diseases.
* Refractory nausea, vomiting, or chronic gastrointestinal diseases, or inability to swallow oral medications
* Hepatic encephalopathy, hepatorenal syndrome, or ≥ Child Pugh B-grade cirrhosis.
* Interstitial lung disease (ILD).
* Serious neurological or mental disorders.
* Active autoimmune diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 762 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Event(s) (AEs) | From Cycle 1 Day 1 (C1D1) to disease progression or death, up to 2 years (each cycle is 14 days).
  An adverse event (AE) is defined as any untoward medical occurrence in a patient and which does not necessarily have a causal relationship with this treatment. Severity is determined according to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0)

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | From Cycle 1 Day 1 (C1D1) to disease progression or death, up to 2 years (each cycle is 14 days).
  Percentage of Participants who Achieve a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR).ORR by the Investigator According to RECIST v1.1
Disease Control Rate (DCR) | From Cycle 1 Day 1 (C1D1) to disease progression or death, up to 2 years (each cycle is 14 days).
  Percentage of Participants who Achieve a BOR of CR, PR, or Stable Disease (SD).DCR by the Investigator According to RECIST v1.1
Time to Response (TTR) | Time from Cycle 1 Day 1 until the date that measurement criteria for CR or PR (whichever is first recorded) are first met, up to 2 years (each cycle is 14 days).
  TTR by the Investigator According to RECIST v1.1
Duration of Response (DOR) | Date of first evidence of CR or PR to date of disease progression or death from any cause, approximately 2 years
  DOR by the Investigator According to RECIST v1.1
Progression-Free Survival (PFS) | Date of first evidence of CR or PR to date of disease progression or death from any cause, approximately 2 years
  PFS by the Investigator According to RECIST v1.1
Overall survival (OS) | Cycle 1 Day 1 to date of death from any cause, up to 5 years (each cycle is 14 days)
  Defined as the time from C1D1 to death from any cause by the Investigator According to RECIST v1.1
Plasma Concentrations of HS-10370 | Cycle 1 Day 1 to date of death from any cause. Various timepoints from Cycle 1 Day 1 through study treatment discontinuation, up to 2 years. (each cycle is 14 days)
  Defined as the time from C1D1 to death from any cause
Maximum plasma concentration (Cmax) | Cycle 1 Day 1 to date of death from any cause, up to 2 years. Various timepoints from Cycle 1 Day 1 through study treatment discontinuation (each cycle is 14 days)
  Cmax is defined as maximum observed serum concentration obtained directly from the observed concentration-time data.
Time of maximum concentration (Tmax) | Cycle 1 Day 1 to date of death from any cause, up to 2 years. Various timepoints from Cycle 1 Day 1 through study treatment discontinuation (each cycle is 14 days)
  Tmax is defined as the time required for a drug to reach peak concentration in plasma.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Sun Yat-sen University Cancer Center, Shanghai